CLINICAL TRIAL: NCT06696833
Title: Assessment of the Safety and Efficacy of Allogeneic CD19-targeted CAR-γδT Cell Infusion Therapy in Relapsed/Refractory B Cell Acute Lymphoblastic Leukemia: A Single-Arm, Open-Label, Prospective Study
Brief Title: Allogeneic CD19-targeted CAR-γδT Cell Infusion Therapy in Relapsed/Refractory B Cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10304-BAL-01
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult
Keywords: B-ALL
MeSH Terms: conditions — Burkitt Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with relapsed/refractory B cell Acute lymphoblastic Leukemia (Experimental): In this study, we adopted a 3+3 design with dose escalation. A conditional chemotherapy regimen of fludarabine and cyclophosphamide will be administered, and each dose group received treatment on Days 0 through i.v. injection, with bone marrow examination performed on Days 14 and 28 to assess tumor burden. Upon assessment by the investigators and discussion with the Safety Review Committee (SRC), it will be determined that whether patients may benefit from additional infusions. With SRC approval, the number of administrations could be increased. At the end of dose escalation, the SRC may decide to adjust the number of participants in the designated dose group as deemed appropriate.
  Interventions: Biological: QH10304-BAL-01; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: QH10304-BAL-01 — dose escalation (3+3) : dose 1 (3 × 10^8cells/kg) ,dose 2 (1 × 10^9 cells/kg) ,dose 3 (3 × 10^9cells/kg)
Drug: Fludarabine — Intravenous fludarabine 30mg/m2 on days-6 to -3,the infusion dose is adjusted according to the subject's condition
Drug: Cyclophosphamide — Intravenous cyclophosphamide 1000mg/m2 on days -5 to -3, the infusion dose is adjusted according to the subject's condition

SUMMARY:
This clinical trial aims to investigate the safety, optimal dosage, and effectiveness of allogeneic CD19-targeted CAR-γδT Cell in treating CD19-positive relapsed/refractory B-ALL

DETAILED DESCRIPTION:
Primary Objective:

To assess the safety of allogeneic CD19-targeted CAR-γδT Cell in the treatment of relapsed/refractory B-ALL, and to determine the recommended dose (RP2D) for the phase II study.

Secondary Objective:

To evaluate the efficacy of allogeneic CD19-targeted CAR-γδT Cell in the treatment of relapsed/refractory B-ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14 years, gender not specified;
2. Diagnosed with B-ALL according to the World Health Organization (WHO) classification of hematopoietic and lymphoid tissue tumors (2022 version);
3. Meet the diagnosis of relapsed/refractory leukemia, excluding isolated extramedullary relapse; For relapsed or refractory B-ALL, including any of the following situations: a) Relapse: Peripheral blood or bone marrow recurrence of primitive cells >5% or extramedullary lesions appear again after complete remission; b) Refractory: Primary refractory patients who fail to achieve complete remission after standard induction chemotherapy；those with positive measurable residual disease can also be included；
4. Flow cytometry confirms positive CD19 expression in leukemia cells；
5. Estimated survival >3 months;
6. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2;
7. The vital organs function in accordance with the following requirements:

   7.1Left ventricular ejection fraction (LVEF) ≥50%; 7.2Pulmonary function：normal oxygen saturation without oxygen supplementation; 7.3Total bilirubin (TBil) ≤3×upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN； 7.4Creatinine ≤1.5×ULN;
8. Pregnancy test must be negative, and fertile non-abstinent female patients must agree to use effective contraception from the start of self-screening to 1 year after cell infusion. Fertile male patients with fertile partners must agree to use effective contraception from the start of self-screening to 1 year after cell infusion, and should not donate semen or sperm throughout the study period；
9. No obvious hereditary diseases；
10. The subject and their legal guardian voluntarily participate in this study, understand the trial information and objectives, and provide informed consent with a signed and dated signature.

Exclusion Criteria:

1. Patients with severe autoimmune diseases or immunodeficiency diseases;
2. Patients with a history of severe central nervous system diseases, such as uncontrolled seizures, stroke, severe brain injury resulting in aphasia, paralysis, dementia, Parkinson's disease, psychiatric disorders, etc.;
3. Any unstable diseases occurring within screening period (including but not limited to): unstable angina, ischemic or cerebrovascular accidents, myocardial infarction, severe arrhythmias requiring drug treatment (such as rapid atrial fibrillation, high-degree atrioventricular block, ventricular tachycardia, ventricular fibrillation, or torsades de pointes), cardiac catheterization or coronary artery stenting, or coronary artery bypass surgery, thrombotic or embolic events.
4. Active graft-versus-host disease requiring continued systemic therapy;
5. The presence of anti-FMC63 and a positive DSA reaction;
6. Patients who have previously received CAR-T cell therapy within 6 months or donor lymphocyte infusion within 6 weeks before screening;
7. History of or concomitant active malignant tumors, excluding cured non-invasive basal cell or squamous cell skin cancer, uterine cervical carcinoma in situ or localized prostate cancer or breast ductal carcinoma in situ without recurrence for at least 2 years;
8. Presence of other severe medical conditions as determined by the investigator, such as uncontrolled hypertension or diabetes, severe renal insufficiency, severe pulmonary dysfunction, etc.;
9. Other severe or persistent active infections;
10. Other conditions deemed by the investigator to potentially increase subject risk or interfere with trial results.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | within 28 days after receiving the infusion
  * Grade ≥ 4 CRS, or Grade 3 CRS that has not resolved to Grade 1 or 2 within 7 days of onset;
  * Grade 4 ICANS or Grade 3 ICANS lasting ≥ 96 hours;
  * Other Grade 3 or higher AEs associated with allogeneic CD19-targeted CAR-γδT Cell and lasting ≥ 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, China, Jiangsu, China